CLINICAL TRIAL: NCT04174599
Title: A Phase III, Multi-Center, Randomized, Open-Label, Active-Controlled Study to Compare the Efficacy and Safety of F-627 and GRAN® in the Prophylactic Treatment for Chemotherapy-Induced Neutropenia
Brief Title: Study to Compare the Efficacy and Safety of F-627 and GRAN®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EVIVE Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP11631
Record Dates: First submitted 2019-07-08; First posted 2019-11-22 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — Filgrastim

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-627 (Experimental): F-627 (20 mg/dose, s.c.) on day 3 of each cycle, i.e., 48 ± 4 h after the start of chemotherapy
  Interventions: Drug: F-627
- GRAN® (Active Comparator): GRAN® [5 μg/kg/day, s.c., once daily (± 4 h) up to 2 weeks or until neutrophil count returns to 5.0 × 10^9/L] on day 3 of each cycle, i.e., 48 ± 4 h after the start of chemotherapy
  Interventions: Drug: GRAN®

INTERVENTIONS:
Drug: F-627 — Day 3 of each cycle, i.e., 48 ± 4 h after starting chemotherapy
  Other Names: Recombinant Human Granulocyte Colony Stimulating Factor-Fc Fusion Protein
  Arms: F-627
Drug: GRAN® — Since day 3 of each cycle, i.e., 48 ± 4 h after starting chemotherapy, continuous treatment for ≤ 2 weeks or until ANC recovers to 5.0 × 10^9/L from nadir (investigators may refer to ANC test results from the Department of Laboratory Medicine of each study sites to decide when to discontinue GRAN®)
  Other Names: Filgrastim
  Arms: GRAN®

SUMMARY:
A Phase III, Multi-Center, Randomized, Open-Label, Active-Controlled Trial to Compare the Efficacy and Safety of Recombinant Human Granulocyte Colony Stimulating Factor-Fc Fusion Protein (F-627) and Recombinant Human Granulocyte Colony Stimulating Factor (GRAN®) in the Prophylactic Treatment for Chemotherapy-Induced Neutropenia

DETAILED DESCRIPTION:
Study Stage: Phase III

Study Population: Female patients with breast cancer will be enrolled to receive at least 4 cycles of Epirubicin + Cyclophosphamide (EC) chemotherapy, that is: epirubicin 100 mg/m^2 and cyclophosphamide 600 mg/m^2.

Study Design: A multi-center, randomized, open-label, active-controlled phase III clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent form and able to comply with protocol requirements;
2. 18-75 years old;
3. Female postoperative patients with breast cancer who require adjuvant chemotherapy, and are planned to receive at least 4 cycles of EC chemotherapy, namely epirubicin 100 mg/m^2 + cyclophosphamide 600 mg/m^2;
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
5. Absolute neutrophil count (ANC) ≥ 2.0 × 10^9/L, hemoglobin (Hb) ≥ 11.0 g/dL, and platelet (PLT) ≥ 100 × 10^9/L prior to enrollment;
6. Hepatic and renal functions: Total bilirubin ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN, serum creatinine ≤ 1.5 × ULN;
7. Left ventricular ejection fraction > 50%;
8. Women without child-bearing potential, i.e., women who have had menopause for at least 1 year or who have undergone sterilization (bilateral tubal ligation, double oophorectomy or hysterectomy); patients with child-bearing potential should agree to take appropriate contraceptive measures, including condoms, spermicidal condoms, foams, gels, contraceptive barrier, intrauterine devices (IUD), and contraceptives (oral or injection), starting from 1 month before the start of the study until 30 days after the end of the study.

Exclusion Criteria:

1. Radiation therapy within 4 weeks prior to enrollment;
2. Patients with breast cancer who have received neoadjuvant chemotherapy before surgery;
3. Prior bone marrow or stem cell transplant;
4. With other malignant tumors other than breast cancer;
5. Patients who have received a treatment with recombinant human granulocyte colony stimulating factor within 6 weeks prior to randomization;
6. Diagnosed with acute congestive heart failure, cardiomyopathy, or myocardial infarction by clinical diagnosis, ECG or other approaches;
7. With any disease that may cause splenomegaly;
8. With acute infection, chronic active Hepatitis B within 1 year (unless patients tested negative for HBsAg prior to enrollment), or Hepatitis C;
9. Women in pregnancy or breastfeeding;
10. Known HIV positive or AIDS;
11. With active tuberculosis (TB); history of TB exposure, unless negative for tuberculin test; TB patients undergoing treatment; or suspected TB evaluated by chest x-ray;
12. With sickle cell anemia;
13. With alcohol or drug abuse that may affect the compliance with the study;
14. With known hypersensitivity to granulocyte colony stimulating factor or excipients;
15. Have received any other investigational drug within 1 month or 5 half-lives of the investigational drugs prior to enrollment (whichever is longer);
16. Patients with diseases or symptoms unsuitable for participating in the trial. For example, the study drugs may compromise the health of the patient or the assessment of adverse events may be affected.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female postoperative patients with breast cancer who require adjuvant chemotherapy, and are planned to receive at least 4 cycles of EC chemotherapy, namely epirubicin 100 mg/m^2 + cyclophosphamide 600 mg/m^2;
Enrollment: 242 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Doctor, Principal Investigator — Fudan University Shanghai Cancer Centre
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang Q, Wang Z, Yao W, Wang S, Zhang G, Chen J, Hou Q, Li S, Li H, Ye C, Sun T, Yang H, Chen Z, Wang Z, Liu X, Geng C, Li X, Zhang J, Zheng H, Shao Z. A randomized, multicenter phase III Study of once-per-cycle administration of efbemalenograstim alfa (F-627), a novel long-acting rhG-CSF, for prophylaxis of chemotherapy-induced neutropenia in patients with breast cancer. BMC Cancer. 2024 Sep 13;24(1):1143. doi: 10.1186/s12885-024-12892-5. PMID 39272058

RESULTS

PARTICIPANT FLOW:
Groups:
- F-627: F-627 (20 mg/dose, s.c.) on day 3 of each cycle, i.e., 48 ± 4 h after the start of chemotherapy
  F-627: Single dose pre-filled syringe
- GRAN®: Recombinant Human Granulocyte Colony Stimulating Factor (GRAN®) [5 μg/kg/day, s.c., once daily (± 4 h) up to 2 weeks or until neutrophil count returns to 5.0 × 10^9/L] on day 3 of each cycle, i.e., 48 ± 4 h after the start of chemotherapy
  GRAN®: Multi-dose pre-filled syringe
Period: Overall Study
Arm/Group | F-627 | GRAN®
Started | 122 (The started participants were all the subjects randomized, but the baseline participants were those randomized subjects received one study drugs at least. A total of 122 subjects were enrolled and randomized in F-627 group. Only 120 randomized patients received one study drugs at least, and included in the full analysis set (FAS), which were consisted of the baseline population.) | 120 (The started participants were all the subjects randomized, but the baseline participants were those randomized subjects received one study drugs at least. A total of 120 subjects were enrolled and randomized in GRAN group. Only 119 randomized patients received one study drugs at least, and included in the full analysis set (FAS), which were consisted of the baseline population.)
Completed | 113 | 101
Not Completed | 9 | 19

BASELINE CHARACTERISTICS:
Population: The started participants were all the subjects randomized, but the baseline participants were those randomized subjects received one study drugs at least.
  A total of 242 subjects were enrolled and randomized. Only 239 randomized patients received one study drugs at least, and included in the full analysis set (FAS), which were consisted of the baseline population.
Groups:
- Total: Total of all reporting groups
Arm/Group | F-627 | GRAN® | Total
Number analyzed (Participants) | 120 | 119 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (9.32) | 48.5 (9.14) | 48.8 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 119 | 239
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 120 | 119 | 239
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 120 | 119 | 239
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 120 | 119 | 239
Height [Mean (Standard Deviation); unit: m] | 157.97 (5.061) | 157.87 (5.524) | 157.92 (5.286)
Weight [Mean (Standard Deviation); unit: kg] | 58.96 (8.945) | 59.24 (8.487) | 59.10 (8.703)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.609 (3.278) | 23.782 (3.336) | 23.695 (3.301)
body surface area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.591 (0.123) | 1.594 (0.116) | 1.593 (0.119)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Grade 3 or 4 Neutropenia (ANC <1.0×10^9/L) in Cycle 1
Description: Grade 3 defined as ANC <1.0×10^9/L and Grade 4 defined as ANC<0.5×10^9/L. According to the study protocol, the outcome measure "Duration of Grade 3 or 4 Neutropenia (days)" applied to all participants with a valid ANC level, rather than those with an ANC level of < 1.0 × 109/L. The value of 0 represents the participant experienced 0 days with Grade 3 or 4 Neutropenia (days). Whereas exclusion of a participant from the analysis indicates a lack of ANC data of the participant.
  The mean value was calculated as the sum of the durations (days) of ANC < 1.0 × 109/L for all participants with valid ANC level (the numerator) divided by the number of participants (the denominator).
Time Frame: Cycle 1, the first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
days | 0.68 (1.100) | 0.71 (0.967)

2. Secondary Outcome: Number of Participants With Grade 3 or 4 Neutropenia in Cycle 1
Description: Grade 3 defined as ANC <1.0×10^9/L and Grade 4 defined as ANC<0.5×10^9/L
Time Frame: Cycle 1, the first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
Participants | 41 | 51

3. Secondary Outcome: Number of Participants With Grade 3 or 4 Neutropenia in Cycle 2
Description: Grade 3 defined as ANC <1.0×10^9/L and Grade 4 defined as ANC<0.5×10^9/L
Time Frame: Cycle 2, the second of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 2
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 117 | 107
Participants | 7 | 7

4. Secondary Outcome: Number of Participants With Grade 3 or 4 Neutropenia in Cycle 3
Description: Grade 3 defined as ANC <1.0×10^9/L and Grade 4 defined as ANC<0.5×10^9/L
Time Frame: Cycle 3, the third of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 3
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 115 | 103
Participants | 4 | 18

5. Secondary Outcome: Number of Participants With Grade 3 or 4 Neutropenia in Cycle 4
Description: Grade 3 defined as ANC <1.0×10^9/L and Grade 4 defined as ANC<0.5×10^9/L
Time Frame: Cycle 4, the last of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 4
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 114 | 101
Participants | 10 | 10

6. Secondary Outcome: Duration of Grade 3 or 4 Neutropenia in Cycle 2
Description: as for outcome 1
Time Frame: Cycle 2, the second of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 117 | 107
days | 0.1 (0.35) | 0.1 (0.25)

7. Secondary Outcome: Duration of Grade 3 or 4 Neutropenia in Cycle 3
Description: as for outcome 1
Time Frame: Cycle 3, the third of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 115 | 103
days | 0.0 (0.18) | 0.2 (0.54)

8. Secondary Outcome: Duration of Grade 3 or 4 Neutropenia in Cycle 4
Description: as for outcome 1
Time Frame: Cycle 4, the last of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 114 | 101
days | 0.1 (0.38) | 0.1 (0.41)

9. Secondary Outcome: Number of Participants With Grade 4 Neutropenia in Cycle 1
Description: Grade 4 neutropenia is defined as ANC < 0.5 × 10^9/L.
Time Frame: Cycle 1, the first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
Participants | 17 | 19

10. Secondary Outcome: Number of Participants With Grade 4 Neutropenia in Cycle 2
Description: Grade 4 neutropenia is defined as ANC < 0.5 × 10^9/L.
Time Frame: Cycle 2, the second of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 2
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 117 | 107
Participants | 2 | 1

11. Secondary Outcome: Number of Participants With Grade 4 Neutropenia in Cycle 3
Description: Grade 4 neutropenia is defined as ANC < 0.5 × 10^9/L.
Time Frame: Cycle 3, the third of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 3
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 115 | 103
Participants | 0 | 4

12. Secondary Outcome: Number of Participants With Grade 4 Neutropenia in Cycle 4
Description: Grade 4 neutropenia is defined as ANC < 0.5 × 10^9/L.
Time Frame: Cycle 4, the last of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 4
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 114 | 101
Participants | 2 | 4

13. Secondary Outcome: Duration of Grade 4 Neutropenia in Cycle 1
Description: Grade 4 neutropenia is defined as ANC < 0.5 × 10^9/L. According to the study protocol, the outcome measure "Duration of Grade 3 or 4 Neutropenia (days)" applied to all participants with a valid ANC level, rather than those with an ANC level of < 1.0 × 109/L. The value of 0 represents the participant experienced 0 days with Grade 3 or 4 Neutropenia (days). Whereas exclusion of a participant from the analysis indicates a lack of ANC data of the participant.
  The mean value was calculated as the sum of the durations (days) of ANC < 1.0 × 109/L for all participants with valid ANC level (the numerator) divided by the number of participants (the denominator).
Time Frame: Cycle 1, the first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
days | 0.3 (0.69) | 0.2 (0.58)

14. Secondary Outcome: Duration of Grade 4 Neutropenia in Cycle 2
Description: as for outcome 13
Time Frame: Cycle 2, the second of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 117 | 107
days | 0.0 (0.13) | 0.0 (0.10)

15. Secondary Outcome: Duration of Grade 4 Neutropenia in Cycle 3
Description: as for outcome 13
Time Frame: Cycle 3, the third of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 115 | 103
days | 0.0 (0.00) | 0.1 (0.34)

16. Secondary Outcome: Duration of Grade 4 Neutropenia in Cycle 4
Description: as for outcome 13
Time Frame: Cycle 4, the last of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 114 | 101
days | 0.0 (0.13) | 0.0 (0.20)

17. Secondary Outcome: Overall Duration of Grade 3 or 4 Neutropenia in 4 Cycles
Description: Grade 3 defined as ANC <1.0×10^9/L and Grade 4 defined as ANC<0.5×10^9/L According to the study protocol, the outcome measure "Duration of Grade 3 or 4 Neutropenia (days)" applied to all participants with a valid ANC level, rather than those with an ANC level of < 1.0 × 109/L. The value of 0 represents the participant experienced 0 days with Grade 3 or 4 Neutropenia (days). Whereas exclusion of a participant from the analysis indicates a lack of ANC data of the participant.
  The mean value was calculated as the sum of the durations (days) of ANC < 1.0 × 109/L for all participants with valid ANC level (the numerator) divided by the number of participants (the denominator).
Time Frame: Overall 4, 21-day chemotherapy cycles(average 12 weeks)
Population: All subjects who have completed cycle 1 at least.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
days | 0.9 (1.44) | 1.1 (1.43)

18. Secondary Outcome: Number of Participants With Grade 2 or Greater Neutropenia in Cycle 1
Description: Grade 2 or greater neutropenia is defined as ANC < 1.5 × 10^9/L
Time Frame: Cycle 1, the first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
Participants | 58 | 67

19. Secondary Outcome: Number of Participants With Grade 2 or Greater Neutropenia in Cycle 2
Description: Grade 2 or greater neutropenia is defined as ANC < 1.5 × 10^9/L
Time Frame: Cycle 2, the second of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 2.
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 117 | 107
Participants | 16 | 14

20. Secondary Outcome: Number of Participants With Grade 2 or Greater Neutropenia in Cycle 3
Description: Grade 2 or greater neutropenia is defined as ANC < 1.5 × 10^9/L
Time Frame: Cycle 3, the third of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 3.
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 115 | 103
Participants | 14 | 30

21. Secondary Outcome: Number of Participants With Grade 2 or Greater Neutropenia in Cycle 4
Description: Grade 2 or greater neutropenia is defined as ANC < 1.5 × 10^9/L
Time Frame: Cycle 4, the last of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 4.
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 114 | 101
Participants | 20 | 26

22. Secondary Outcome: Duration (Days) of Grade 2 or Greater Neutropenia in Cycle 1
Description: Grade 2 or greater neutropenia is defined as ANC < 1.5 × 10^9/L. According to the study protocol, the outcome measure "Duration of Grade 3 or 4 Neutropenia (days)" applied to all participants with a valid ANC level, rather than those with an ANC level of < 1.0 × 109/L. The value of 0 represents the participant experienced 0 days with Grade 3 or 4 Neutropenia (days). Whereas exclusion of a participant from the analysis indicates a lack of ANC data of the participant.
  The mean value was calculated as the sum of the durations (days) of ANC < 1.0 × 109/L for all participants with valid ANC level (the numerator) divided by the number of participants (the denominator).
Time Frame: Cycle 1, the first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 1.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
days | 1.1 (1.30) | 1.0 (1.10)

23. Secondary Outcome: Duration (Days) of Grade 2 or Greater Neutropenia in Cycle 2
Description: as for outcome 22
Time Frame: Cycle 2, the second of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 117 | 107
days | 0.2 (0.50) | 0.2 (0.50)

24. Secondary Outcome: Duration (Days) of Grade 2 or Greater Neutropenia in Cycle 3
Description: as for outcome 22
Time Frame: Cycle 3, the third of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 3.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 115 | 103
days | 0.1 (0.42) | 0.4 (0.67)

25. Secondary Outcome: Duration (Days) of Grade 2 or Greater Neutropenia in Cycle 4
Description: as for outcome 22
Time Frame: Cycle 4, the last of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 4.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 114 | 101
days | 0.3 (0.68) | 0.3 (0.63)

26. Secondary Outcome: The Absolute Neutrophil Counts (ANC) Nadir From Day 3 to Day 13 of Cycle 1
Description: The minimum value of ANC measured from day 3 to day 13 of cycle 1
Time Frame: From day 3 to day 13 of cycle 1 (11 days)
Population: All subjects who have completed cycle 1
Measure: Mean (Standard Deviation); unit: 10^9 cell/L
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
10^9 cell/L | 2.058 (1.503) | 1.597 (1.197)

27. Secondary Outcome: Number of Participants With Febrile Neutropenia (FN) in Cycle 1
Description: FN is defined as ANC < 1.0 × 10^9/L with fever (a single measurement of body temperature >38.3 °C or body temperature ≥ 38.0 °C for more than 1 hr).
Time Frame: Cycle 1, the first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
Participants | 1 | 2

28. Secondary Outcome: Time (Days) of ANC Nadir Recovers to 2.0 × 10^9/L in Cycle 1
Description: If the ANC nadir during the first 13 days of the cycle is < 2.0 × 10^9/L, the recovery time = ((date of ANC ≥ 2.0 ×10^9/L) - (date of ANC reaching nadir within the cycle) + 1). If the ANC nadir in the first 13 days of the cycle is ≥2.0 × 10^9/L, then the recovery time = 0 days.
Time Frame: Cycle 1, the first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 120 | 119
days | 0.9 (1.01) | 1.0 (0.84)

29. Secondary Outcome: Time (Days) of ANC Nadir Recovers to 2.0 × 10^9/L in Cycle 2
Description: as for outcome 28
Time Frame: Cycle 2, the second of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 117 | 107
days | 0.5 (1.10) | 0.7 (0.99)

30. Secondary Outcome: Time (Days) of ANC Nadir Recovers to 2.0 × 10^9/L in Cycle 3
Description: as for outcome 28
Time Frame: Cycle 3, the third of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 115 | 103
days | 0.4 (0.87) | 0.9 (1.50)

31. Secondary Outcome: Time (Days) of ANC Nadir Recovers to 2.0 × 10^9/L in Cycle 4
Description: as for outcome 28
Time Frame: Cycle 4, the last of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: All subjects who have completed cycle 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | GRAN®
Number analyzed (Participants) | 114 | 101
days | 0.7 (1.14) | 1.2 (1.73)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are recorded from randomization until 30 days after the last dose of the study drug, including AEs that occurred prior to the randomization and worsened during the treatment period, e.g.average 95 days.
Arm/Group | F-627 | GRAN®
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/119
Serious Adverse Events (participants affected / at risk) | 6/120 | 8/119
Other Adverse Events (participants affected / at risk) | 119/120 | 119/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-627 (N=120) | GRAN® (N=119)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (3)
Platelet count decreased (Investigations) | 3 (3) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-627 (N=120) | GRAN® (N=119)
Nausea (Gastrointestinal disorders) | 104 (104) | 102 (102)
Vomiting (Gastrointestinal disorders) | 76 (76) | 89 (89)
Constipation (Gastrointestinal disorders) | 17 (17) | 17 (17)
Abdominal distension (Gastrointestinal disorders) | 14 (14) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 8 (8)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 6 (6)
White blood cell count decreased (Investigations) | 79 (79) | 99 (99)
Neutrophil count decreased (Investigations) | 71 (71) | 99 (99)
Platelet count decreased (Investigations) | 56 (56) | 40 (40)
Alanine aminotransferase increased (Investigations) | 36 (36) | 19 (19)
Aspartate aminotransferase increased (Investigations) | 30 (30) | 14 (14)
Weight decreased (Investigations) | 6 (6) | 7 (7)
Weight increased (Investigations) | 9 (9) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 93 (93) | 83 (83)
Anaemia (Blood and lymphatic system disorders) | 81 (81) | 79 (79)
Bone pain (Musculoskeletal and connective tissue disorders) | 30 (30) | 40 (40)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (19) | 28 (28)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8)
Asthenia (General disorders) | 42 (42) | 35 (35)
Chest discomfort (General disorders) | 8 (8) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 29 (29) | 30 (30)
Dizziness (Nervous system disorders) | 8 (8) | 14 (14)
Headache (Nervous system disorders) | 7 (7) | 15 (15)
Somnolence (Nervous system disorders) | 9 (9) | 4 (4)
Poor quality sleep (Nervous system disorders) | 1 (1) | 7 (7)
Vertigo (Ear and labyrinth disorders) | 27 (27) | 21 (21)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 16 (16)
Insomnia (Psychiatric disorders) | 14 (14) | 16 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7)
Palpitations (Cardiac disorders) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT04174599/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT04174599/SAP_001.pdf